CLINICAL TRIAL: NCT02917447
Title: Evaluation of Web-Based CBT for Women Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-021-13SB; IK2CX000867-01 (NIH)
Record Dates: First submitted 2016-09-23; First posted 2016-09-28 (Estimated); Results first posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: PTSD
Keywords: PTSD; Women Veterans; Online intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DESTRESS-WV (Experimental): Tailored online intervention for PTSD for women Veterans with coach support.
  Interventions: Behavioral: DESTRESS-WV
- Phone Monitoring (Placebo Comparator): Weekly check-in calls from a study coach.
  Interventions: Behavioral: Phone Monitoring

INTERVENTIONS:
Behavioral: DESTRESS-WV — This is an online intervention for PTSD tailored for women Veterans. The intervention is based on cognitive behavioral therapy (CBT). The goal of CBT is to help people recognize and address their thoughts and behaviors in positive ways with the aim of improving their ability to function as well as possible in their lives. Participants will be asked to log on to the website twice per week for about 30-60 minutes each time. Homework assignments will include stress management skills that participants will be asked to practice and apply. A study coach will call each participant once a week for 8 weeks for about 15 minutes to review their progress with the program.
  Arms: DESTRESS-WV
Behavioral: Phone Monitoring — A study coach will call participants once a week for 8 weeks for approximately 15 minutes. The coach will assess participants' PTSD symptoms and safety. She will encourage participants to use the time on the call to discuss any current life issues or problems that they would like. Active listening and rephrasing will be used, while teaching cognitive-behavioral strategies will be avoided.
  Arms: Phone Monitoring

SUMMARY:
The purpose of this study is to evaluate an online PTSD intervention that was adapted for women Veterans, called DElivery of Self TRaining and Education for Stressful Situations-Women Veterans version (DESTRESS-WV). The intervention consists of structured online sessions as well as weekly brief phone calls for additional support with a study coach. Women Veterans with PTSD who are eligible will be randomized to receive either DESTRESS-WV or phone monitoring only for 8 weeks. Participants will be assessed immediately post-treatment as well as at 12 and 24 weeks post-treatment. Investigators hypothesize that participants randomly assigned to DESTRESS-WV will have a greater decrease in severity of PTSD symptoms compared to those randomly assigned to phone monitoring only.

DETAILED DESCRIPTION:
The RCT will target women Veterans with PTSD to compare the adapted, web-based intervention to phone monitoring only. Participants will include women Veterans with PTSD who are not actively receiving PTSD treatment. They will be interviewed via phone for an initial phone screening and eligibility interview and will complete additional online surveys at baseline, post-treatment, and 12-, and 24-week follow-up.

Recruitment. Women Veterans who live in Pacific or Mountain Time Zones with an ICD code for PTSD or a positive VA mandated PTSD screen, with no mental health stop-code in the last 2 months, and who are not on the high risk list for imminent danger to self or others, will be identified using a VINCI data pull. Individuals with these criteria will be mailed up to two invitation letters and a brochure describing the study inviting them to contact the study office. If women do not contact the study office to opt out of the study, the investigators may call them to follow-up. The investigators aim to obtain a sample of 100 individuals that meet study inclusion/exclusion criteria after providing informed consent. Because the investigators aim to recruit participants for approximately 24 months, the investigators will aim to enroll and randomize 4-5 participants per month.

Procedure. The RCT will involve four assessment phases: initial phone screen to ascertain interest and basic inclusion/exclusion eligibility, assessment of diagnostic eligibility in a full eligibility interview, baseline survey of outcomes of interest prior to initiating treatment, and three follow-up surveys of outcomes of interest at post-treatment and 12- and 24-weeks post-treatment. Patients will be randomized to condition following completion of the baseline online survey. The eligibility interview and study coach phone calls will be audio-recorded to ensure adherence to the study protocol.

Phone screen (10-15 minutes). When interested women Veterans contact the study office, study personnel will provide an overview of the study and, for those still interested, conduct an initial pre-consent screening. The purpose of the pre-consent eligibility screening is to quickly determine which candidates are most likely to qualify, thus eliminating the need to conduct consent and full eligibility interviews for those who are unlikely to meet study criteria. If patients are found to be eligible following the pre-consent eligibility screening, study staff will review the consent process, including willingness to be audio-taped during assessments and study coach calls, answer any questions, and mail the consent form to the participant to obtain written consent, along with a demographic form and Life Events Checklist. The full eligibility interview will be scheduled at this time but will only be conducted if and when the signed, written informed consent, HIPAA form, demographic form, and Life Events Checklist have been received in the study office.

Eligibility interview (95-150 minutes). Study personnel will call the potential study participant to conduct the eligibility interview over the phone after written, informed consent has been received in the study office. The interview will assess current PTSD as addressed by the CAPS interview as well as various exclusion criteria. During the course of the interview, if study personnel are concerned about the fit of the study for the potential participant, they will discuss with the PI. Potential participants who are of concern and may show a high risk profile (e.g., multiple past suicide attempts, inpatient hospitalizations, lifetime psychotic disorders) or prominent disorganization while on the phone will be discussed by the PI and co-investigator Dr. Simpson for possible exclusion.

Respondents who do not meet eligibility criteria will be offered a resource list, referred for treatment, and/or be further assessed for suicidality as appropriate. For those who are eligible, contact information (e.g., address, telephone number) and contact information for at least one friend or family member who typically would know the whereabouts of the participant should study staff have difficulty making contact will be recorded. Eligible patients will be invited to complete a baseline online survey.

Baseline and follow-up online surveys (60-90 minutes). The baseline and follow-up surveys (at post-treatment and 12- and 24-week follow-ups) consist of an online survey. Each online survey takes 60-90 minutes to complete. Participants will be compensated for the baseline survey, for each of the follow-up surveys, and a bonus for completing all surveys. If the interval between the eligibility interview and baseline survey is longer than four weeks, we will require re-administration of CAPS via telephone to ensure PTSD status. Participants will be given one-week and one-day reminders to complete the survey. Following completion of the baseline survey, participants will be randomly assigned to one of the conditions.

Randomization scheme. Fifty participants will be randomized to the adapted, web-based intervention and 50 to phone monitoring only. Participants will be randomized following their completion of the baseline survey. Stratification of randomization by rural status will be done to facilitate exploratory analyses of the impact of this variable on trial outcomes. Following randomization, the study coach will arrange an initial telephone session with each participant.

Study conditions. The treatment phase for both study conditions will last 8 weeks; however, participants will have up to 12 weeks to complete the intervention and complete study coach calls, if needed.

Phone monitoring condition. Participants randomized to the phone monitoring condition will receive calls from a study coach once a week for 8 weeks for approximately 10-15 minutes. The coach will assess their PTSD symptoms and safety.

DESTRESS-WV. Those randomly assigned to the web-based intervention will also receive calls from a study coach once a week for 8 weeks to assess PTSD symptoms and safety; the coach will also review the participant's progress with the DESTRESS-WV website. Participants will be instructed to log-on to the website twice per week, with each session taking approximately 30-60 minutes. The web-based intervention consists of 16 sessions involving structured, cognitive-behavioral components, including cognitive restructuring and in-vivo and imaginal exposure. Participants will be reminded of the study office phone number as well as the Veterans Crisis Line phone number at every logon.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* female
* Veteran of the US military
* current PTSD
* reports routine access to computer and Internet
* willing to provide at least one collateral contact
* willing to allow investigators to leave phone messages pertaining to the study
* willing to be audio-taped during assessments and study coach calls

Exclusion Criteria:

* actively engaged in individual therapy in the past two months, or receiving couple's or group therapy in the past two months that focuses on PTSD
* scheduled to receive a future individual therapy appointment or future couples' or group therapy appointment focused on PTSD at a frequency of once per month or more
* active suicidal or violent ideation within the past two months or on the VA "high risk" list for imminent danger to self or others
* moderate or extreme substance use disorder in the past year
* acute psychosis, psychotic episode, or psychotic disorder diagnosis within the past year
* unstable administration schedule or dosing of any antidepressant, anxiolytic, or sedative-hypnotic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is focused on cisgender women.
Enrollment: 102 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keren Lehavot, PhD MS BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehavot K, Litz B, Millard SP, Hamilton AB, Sadler A, Simpson T. Study adaptation, design, and methods of a web-based PTSD intervention for women Veterans. Contemp Clin Trials. 2017 Feb;53:68-79. doi: 10.1016/j.cct.2016.12.002. Epub 2016 Dec 8. PMID 27940187
- [Background] Engel CC, Litz B, Magruder KM, Harper E, Gore K, Stein N, Yeager D, Liu X, Coe TR. Delivery of self training and education for stressful situations (DESTRESS-PC): a randomized trial of nurse assisted online self-management for PTSD in primary care. Gen Hosp Psychiatry. 2015 Jul-Aug;37(4):323-8. doi: 10.1016/j.genhosppsych.2015.04.007. Epub 2015 Apr 13. PMID 25929985
- [Background] Litz BT, Engel CC, Bryant RA, Papa A. A randomized, controlled proof-of-concept trial of an Internet-based, therapist-assisted self-management treatment for posttraumatic stress disorder. Am J Psychiatry. 2007 Nov;164(11):1676-83. doi: 10.1176/appi.ajp.2007.06122057. PMID 17974932
- [Result] Lehavot K, Katon JG, Chen JA, Fortney JC, Simpson TL. Post-traumatic Stress Disorder by Gender and Veteran Status. Am J Prev Med. 2018 Jan;54(1):e1-e9. doi: 10.1016/j.amepre.2017.09.008. PMID 29254558
- [Derived] Chen JA, Shofer J, Barnes ML, Livingston WS, Upham M, Simpson TL. Military Sexual Trauma As a Risk Factor for Treatment Non-Response from an Online, Self-Management Posttraumatic Stress Disorder Treatment for Women Veterans. J Interpers Violence. 2024 May;39(9-10):2214-2237. doi: 10.1177/08862605231216722. Epub 2023 Dec 11. PMID 38073465
- [Derived] Simon N, Robertson L, Lewis C, Roberts NP, Bethell A, Dawson S, Bisson JI. Internet-based cognitive and behavioural therapies for post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2021 May 20;5(5):CD011710. doi: 10.1002/14651858.CD011710.pub3. PMID 34015141
- [Derived] Lehavot K, Millard SP, Thomas RM, Yantsides K, Upham M, Beckman K, Hamilton AB, Sadler A, Litz B, Simpson T. A randomized trial of an online, coach-assisted self-management PTSD intervention tailored for women veterans. J Consult Clin Psychol. 2021 Feb;89(2):134-142. doi: 10.1037/ccp0000556. PMID 33705169

RESULTS

PARTICIPANT FLOW:
Groups:
- DESTRESS-WV: Tailored online intervention for PTSD for women Veterans with coach support.
  DESTRESS-WV: This is an online intervention for PTSD tailored for women Veterans with weekly, 15-minute coach calls. The intervention is based on cognitive behavioral therapy (CBT). The goal of CBT is to help people recognize and address their thoughts and behaviors in positive ways with the aim of improving their ability to function as well as possible in their lives.
  Participants will be asked to log on to the website twice per week for about 30-60 minutes each time. On two occasions, participants will be asked to write about current stressors or hassles. Additionally, on two occasions participants will be asked to write about a traumatic experience and then rewrite it. Participants will be guided in using various coping skills taught in the program during this writing process. Homework assignments will include stress mana
Period: Overall Study
Arm/Group | DESTRESS-WV | Phone Monitoring
Started | 51 | 51
Completed | 44 | 48
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DESTRESS-WV | Phone Monitoring | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (11.3) | 48.9 (12.2) | 49.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 51 | 102
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 49 | 42 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 8 | 14
  White | 36 | 34 | 70
  More than one race | 3 | 6 | 9
  Unknown or Not Reported | 2 | 1 | 3
PTSD Symptom-Checklist -Version 5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — total severity score ranging from 0-80, with higher scores representing greater symptom severity
  units on a scale | 45.8 (10.6) | 45.0 (11.7) | 45.4 (11.1)
Patient Health Questionnaire (PHQ)-8 [Mean (Standard Deviation); unit: units on a scale] — range from 0-24, with a score of 10 or greater indicating major depression
  units on a scale | 13.6 (4.9) | 13.2 (5.5) | 13.4 (5.2)
The Quality of Life (QoL) Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) [Mean (Standard Deviation); unit: units on a scale] — scale ranging from 0-100, with higher scores indicating greater quality of life
  units on a scale | 44.9 (15.5) | 45.5 (12.2) | 45.2 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Checklist (PCL-5)
Description: The PTSD Symptom-Checklist -Version 5 (PCL-5) is a 20-item, self-report instrument that assesses the presence and severity of DSM-V PTSD symptoms in the last month. It was summed for a total severity score ranging from 0-80, with higher scores representing greater symptom severity. Changes from baseline at three separate times post-baseline are reported for each treatment group. These calculations are based on marginal means estimated from a linear mixed model analysis with PCL as the dependent variable; rural status, MST history, study assessment, treatment group, and study assessment by treatment group interaction as the independent fixed effects; and study participant as a random effect.
Time Frame: Baseline, Post-treatment (8-12 weeks after baseline), 3-months post-treatment, 6-months post-treatment
Population: Intent to treat population (all participants assigned to DESTRESS-WV or Phone Monitoring). Linear mixed effects regressions of PCL on categorical follow-up time, adjusted for rural/urban status and MST.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DESTRESS-WV | Phone Monitoring
Number analyzed (Participants) | 51 | 51
units on a scale
  Post - Baseline | -13.1 (2.1) | -8.9 (2.0)
  3-month - Baseline | -13.8 (2.1) | -7.5 (2.0)
  6-month - Baseline | -11.4 (2.1) | -8.9 (2.0)
Statistical Analysis 1: Comparison: DESTRESS-WV vs Phone Monitoring; Test type: Superiority; p = 0.15, Mixed Models Analysis — Omnibus test for difference in change from baseline in PCL by treatment group across the three post-treatment assessments, adjusted for rural/urban status and MST; Fixed effects were study assessment, group, the assessment by group interaction, and covariates. Participant was modeled as a random effect

2. Secondary Outcome: Change in Patient Health Questionnaire-8 (PHQ-8)
Description: The Patient Health Questionnaire-8 (PHQ-8) is a brief self-report assessment of common mental disorders and was used to assess symptoms of depression. The eight items specifically correspond to symptom-based diagnostic criteria in DSM-IV and are summed for a range from 0-24, with a score of 10 or greater indicating major depression. Changes from baseline at three separate times post-baseline are reported for each treatment group. These calculations are based on marginal means estimated from a linear mixed model analysis with PHQ-8 as the dependent variable; rural status, MST history, study assessment, treatment group, and study assessment by treatment group interaction as the independent fixed effects; and study participant as a random effect.
Time Frame: Baseline, Post-treatment (8-12 weeks after baseline), 3-months post-treatment, 6-months post-treatment
Population: Intent to treat population (enrolled in DESTRESS-WV or Phone Monitoring).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DESTRESS-WV | Phone Monitoring
Number analyzed (Participants) | 51 | 51
units on a scale
  Post - Baseline | -3.8 (0.8) | -2.6 (0.7)
  3 month - Baseline | -3.5 (0.8) | -0.6 (0.7)
  6 month - Baseline | -2.3 (0.8) | -1.2 (0.7)
Statistical Analysis 1: Comparison: DESTRESS-WV vs Phone Monitoring; Test type: Superiority; p = .049, Mixed Models Analysis — Omnibus test for difference in change from baseline in outcome by treatment group across the three post-treatment assessments, adjusted for rural/urban status and MST; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Change in the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form
Description: The Quality of Life (QoL) Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) was used to assess quality of life. It consists of 16 items that are summed and transformed to a scale ranging from 0-100, with higher scores indicating greater quality of life. Changes from baseline at three separate times post-baseline are reported for each treatment group. These calculations are based on marginal means estimated from a linear mixed model analysis with QoL as the dependent variable; rural status, MST history, study assessment, treatment group, and study assessment by treatment group interaction as the independent fixed effects; and study participant as a random effect.
Time Frame: Baseline, Post-treatment (8-12 weeks after baseline), 3-months post-treatment, 6-months post-treatment
Population: Intent to treat population (all participants enrolled in DESTRESS-WV or Phone Monitoring).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | DESTRESS-WV | Phone Monitoring
Number analyzed (Participants) | 51 | 51
units on a scale
  Post - Baseline | 9.1 (2.2) | 7.9 (2.1)
  3 month - Baseline | 4.3 (2.2) | 4.8 (2.1)
  6 month - Baseline | 3.0 (2.2) | 3.8 (2.1)
Statistical Analysis 1: Comparison: DESTRESS-WV vs Phone Monitoring; Test type: Superiority; p = 0.92, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected up through the 6-month post-treatment assessment. Adverse Events are reported if they occurred after randomization to study condition.
Description: Hospitalizations were assessed systematically at all assessments. If the reason for the hospitalization was unknown, it is categorized under "general disorders." Symptom exacerbations were defined as an increase of 7 or more points on a shortened-PCL from baseline, assessed during weekly coaching calls during the treatment phase. Statements of hopelessness, suicidal ideation, and ER visits were not systematically assessed in self-report forms but addressed verbally during calls with study staff.
Arm/Group | DESTRESS-WV | Phone Monitoring
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/51
Serious Adverse Events (participants affected / at risk) | 7/51 | 5/51
Other Adverse Events (participants affected / at risk) | 14/51 | 16/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DESTRESS-WV (N=51) | Phone Monitoring (N=51)
Hospitalizations (General disorders) | 2 (3) | 2 (3)
Hospitalizations (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalizations (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalizations (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalizations (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalizations (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Hospitalizations (Psychiatric disorders) | 0 (0) | 1 (1)
Hospitalizations (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DESTRESS-WV (N=51) | Phone Monitoring (N=51)
Symptom exacerbation (Psychiatric disorders) | 7 (12) | 7 (9) — Symptom exacerbations were defined as an increase of 7 or more points on a shortened-PCL from baseline, assessed during every weekly coaching call during the treatment phase.
Emergency Room Visit (General disorders) | 4 (4) | 4 (4)
Hopelessness (Psychiatric disorders) | 2 (2) | 3 (4) — Participant reported hopelessness during weekly coaching call.
Suicidal ideation (Psychiatric disorders) | 1 (1) | 4 (6) — Participant reported suicidal ideation during contact with study staff.
Distress (Psychiatric disorders) | 1 (1) | 2 (2) — Participant reported distress related to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT02917447/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT02917447/Prot_SAP_001.pdf